CLINICAL TRIAL: NCT05087420
Title: Migraine in Poland - a Web-based Cross-sectional Survey
Acronym: MIGinPOL2021
Status: Completed | Type: Observational
Sponsor: Swiat Zdrowia (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Marcin Straburzynski, General practitioner, Swiat Zdrowia
Other Study IDs: MIGinPOL2021
Record Dates: First submitted 2021-09-19; First posted 2021-10-21 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Migraine
Keywords: migraine; headache; rhinosinusitis; COVID-19
MeSH Terms: conditions — Migraine Disorders; Headache; Rhinosinusitis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A survey of Polish respondents will aim to define migraine characteristics in Polish subjects. To achieve this, a structured questionnaire based mainly on American Migraine Prevalence and Prevention Study has been prepared to serve as a tool for data extraction. The obtained data should allow for defining disease parameters, burden and received treatments. Additionally questions regarding patients rhinological symptoms and COVID-19-related history were included.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate in the study

Exclusion Criteria:

* responses missing in questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participant will be recruited from miscellaneous sources including: specialist headache practices, primary care clinics, patients associations. An invitation would be also extended via social and traditional media and employers.
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Headache phenotype | in the preceding year
  Classification of reported headache according to International Classification of Headache Disorders
Migraine burden | in the preceding year
  Consequences of the disease measured by the Migraine Disability Assessment Test

SECONDARY OUTCOMES:
Monthly headache days | in the preceding month
  Number of days per month
Monthly headache days | in the preceding year
  Number of days per year
Time from last headache professional consultation | in the preceding 10 years
  Number of months
Migraine diagnosed by headache professional | in the preceding 10 years
  yes/no
Age at diagnosis | from the onset of headache (time frame up to 99 years)
  years
Comoribidities | in the preceding year
  Disease according to International Classsification of Disease 10
Type of previous headache professional consultation | in the preceding 10 years
  Name of headache profession/speciality
Number of consultations in the last year | in the last 12 months
  Number 0-100
Number of consultations in the last year because of headaches | in the last 12 months
  Number 0-100
Number of days spent in hospital in the last year because of headaches | in the last 12 months
  Number 0-100
Acute treatment used | in the preceding 10 years
  Name of abortive medication
Preventive treatment used | in the preceding 10 years
  Name of abortive medication
Acute treatment frequency | in the last 3 months
  Number of days per month
Preventive treatment frequency | in the last 12 months
  Number of months form the last dose
Preventive treatment effectiveness | in the last 12 months
  Likert scale
Employment | in the last 12 months
  Type of employment
Time spent at work | in the last 12 months
  Number of hours per week
Work absence due to headache | in the last month
  Number of days per month
Presenteeism | in the last month
  Number of days per month
PHQ-9 Patient Health Questionnaire | in the last 2 weeks
  Number
Sinus headache | in the last 3 months
  Number of days
Sinonasal symptoms accompanying headache | in the last 12 months
  Type of symptoms
Sinonasal symptoms not associated with headache | in the last 12 months
  Type of symptom
COVID-19 association with headache | in the last 2 years
  Likert scale
COVID-19 vaccine association with headache | in the last year
  Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Marta Waliszewska-Prosół, MD, PhD, Study Chair — Departament of Neurolog, Wrocław Medical University
Locations (2):
- Poland (2):
  - Marcin Straburzyński, Dźwierzuty, Warmian-Masurian Voivodeship
  - Department of Neurology, Wrocław Medical University, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straburzynski M, Waliszewska-Prosol M, Nowaczewska M, Czapinska-Ciepiela EK, Gryglas-Dworak A, Budrewicz S. Prevalence of cranial autonomic symptoms in frequent episodic tension-type headache: A post hoc analysis of the cross-sectional Migraine in Poland study. Dent Med Probl. 2024 Jul-Aug;61(4):489-493. doi: 10.17219/dmp/175611. PMID 38652923